CLINICAL TRIAL: NCT06056570
Title: A Phase 1B Open Label Evaluation of the PK and PD of Dotinurad and Drug-Drug Interaction of Dotinurad and Allopurinol in U.S. Patients with Gout and Hyperuricemia
Brief Title: Open Label PK, PD and DDI of Dotinurad and Allopurinol in Gout Patients with Hyperuricemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Urica Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UR1-DOT-103
Record Dates: First submitted 2023-09-07; First posted 2023-09-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — dotinurad; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dotinurad 2mg (Experimental): dotinurad 2mg q.d.
  Interventions: Drug: dontinurad; Drug: dotinurad + allopurinol; Drug: allopurinol
- dotinurad 4mg (Experimental): dotinurad 4mg q.d.
  Interventions: Drug: dontinurad; Drug: dotinurad + allopurinol; Drug: allopurinol

INTERVENTIONS:
Drug: dontinurad — dotinurad alone
Drug: dotinurad + allopurinol — dotinurad + allopurinol 300mg
Drug: allopurinol — allopurinol 300 mg alone

SUMMARY:
A open label multi-center 3-period multidose, PK/PD and drug-drug interaction (DDI) study to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of 7 days of treatment with two doses of dotinurad monotherapy, and to evaluate the effect of dotinurad, as monotherapy and in combination with allopurinol, versus allopurinol monotherapy, on the PK of each, and to assess the additive PD effects on serum uric acid and urinary urate excretion in U.S. patients with gout and hyperuricemia

ELIGIBILITY:
Inclusion Criteria:

* 1. In the opinion of the investigator, the patient is capable of understanding and complying with protocol requirements.

  2. Patients with a diagnosis of gout based on American College of Rheumatology criteria (1997). Patients must fulfill at least 3 of the following, with one of those 3 being (i) hyperuricemia.
  1. More than one attack of acute arthritis
  2. Maximum inflammation developed within 1 day
  3. Monoarthritis attack
  4. Redness observed over joints
  5. First metatarsophalangeal joint painful or swollen
  6. Unilateral first metatarsophalangeal joint attack
  7. Unilateral tarsal joint attack
  8. Tophus (proven or suspected)
  9. Hyperuricemia.
  10. Asymmetric swelling within a joint on x-ray
  11. Subcortical cysts without erosions on x-ray
  12. Monosodium urate monohydrate microcrystals on joint fluid during attack
  13. Joint fluid culture negative for organisms during attack 3. The patient signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a patient fast for any laboratory evaluations.

      4. Negative COVID-19 test by either PCR or rapid antigen test at screening and check-in prior to first period, and agrees to be compliant with all COVID-19 measures mandated by the CRU prior to screening/entry into the trial.

      5. Male or female between 18 and 75 years of age (inclusive). To be eligible, females can be either of NCBP (confirmed by surgical history, medical history of twelve consecutive months of amenorrhea, or FSH levels) or females of childbearing potential must be on a reliable method of birth control and also have a negative urine human chorionic gonadotropin (hCG) pregnancy test results on the Study Day -1.

      6. Screening serum uric acid level of ≥7 mg/dl.

  a. If a patient is not on uric acid-lowering therapies (ULT) prior to screening, the required fasting sUA level is at least one ≥7 mg/dl during Screening b. If a patient is on ULT prior to screening, the required fasting sUA level is at least one =>7 mg/dl between Day -7 and Day -1 7. Screening liver enzymes (LFTs) <1.5x ULN. Total bilirubin <1x ULN. For patients with documented Gilbert Syndrome, total bilirubin ≤3 x ULN with direct bilirubin <1x ULN.

  8. Screening renal function eGFR ≥ 60 mL/min/1.73m2. 9. Pre-dose hemoglobin should be within the normal range. 10. Body mass index (BMI) ≥ 18.5 and ≤ 40.0 (kg/m2) and a body weight of no less than 50 kg.

  11. Medically healthy with no clinically significant screening results including but not limited to:
  1. Laboratory profiles other than sUA
  2. Urinalysis
  3. Vital signs
  4. Electrocardiograms (ECGs)
  5. Physical examination 12. No use of tobacco or nicotine containing products (including smoking cessation products), for a minimum of 3 months prior to dosing.

     Exclusion Criteria:
* 1. The subject has current or historical evidence of any clinically significant disease or condition that might complicate the subject's participation, or, in the opinion of the Investigator, may place the subject at an unacceptable risk as a participant in this trial, may interfere with the interpretation of safety and/or tolerability data obtained in the trial, or may interfere with the absorption, distribution, metabolism, or excretion of the study drug.

  2. Patients with unstable angina, New York Heart Association Class III or IV heart failure, myocardial infarction, stroke, or deep venous thrombosis within 1 year prior to Day 1.

  3. QT interval corrected for heart rate according to Fridericia's formula >470 msec in females and >450 msec in males during Screening, confirmed by a repeat assessment.

  4. History of or presence of kidney stones. 5. History of or presence of malignancy in the last 5 years other than treated cutaneous basal or squamous cell carcinoma.

  6. Urological disorder not well controlled. 7. Peptic ulcer disease requiring active treatment. 8. Cannot safely discontinue uric acid-lowering medication 14 days prior to study start to 9 days after the last dose of study medication was administered.

  9. Surgery within the past 90 days prior to dosing as determined by the Principal Investigator to be clinically relevant.

  10. Use of agents that could confound serum uric acid analysis (eg, long-term use of salicylates >100 mg or use of losartan).

  11. Patients with an acute gout flare during the screening period that had not resolved 1 week prior to the first dose of study.

  12. Hypersensitivity or intolerance to allopurinol, dotinurad or colchicine. 13. Positive for HLA-B*58:01 allele 14. History or presence of alcoholism or chronic drug abuse within the past 2 years.

  15. Psychiatric disorder or social situation that prevents compliance with the protocol.

  16. Female patients who are pregnant or lactating. 17. Positive results for the urine drug /alcohol breath test/cotinine at check-in.

  18. Positive results at screening for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), Hepatitis C antibodies (HCV).

  19. Patient's semi-recumbent blood pressure is less than 90/40 mmHg or greater than 155/90 mmHg during Screening and Day -1.

  20. Stable dose of medications for long-term conditions such as diabetes, high cholesterol, hypertension, asthma, etc. are allowed (provided that the patient has been on a stable dose for at least 30 days prior to Screening and is not expected to require dose adjustment during the study through 7 days post study).

  21. Patient reports receiving a strong or moderate inhibitor of CYP3A4 or a P-gp inhibitor within 1 month prior to study drug dosing, due to potential interactions with colchicine.

  22. Patient has taken azathioprine, Imuran, or other medications that may interact with allopurinol within 1 month prior to study drug dosing 23. Participation in another clinical trial within 30 days of last IP administration or 5 half-lives (whichever is longer) of administration of any study drug evaluated in that trial prior to screening for this trial. Previous participation in a dotinurad trial is also exclusionary.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentrations (Cmax) | 7 days
  To evaluate the Cmax of dotinurad 2mg, dotinturad 4mg, and allopurinol 300mg
Area under the plasma concentration versus time curve (AUC) | 7 days
  To evaluate the AUC of dotinurad 2mg, dotinturad 4mg, and allopurinol 300mg
Time to maximum plasma concentration (Tmax) | 7 days
  To evaluate the Tmax of dotinurad 2mg, dotinturad 4mg, and allopurinol 300mg
Terminal half life (T1/2) | 7 days
  To evaluate the T1/2 of dotinurad 2mg, dotinturad 4mg, and allopurinol 300mg

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Research of West Florida, Clearwater, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Southwest Rheumatology Research, Mesquite, Texas
  - Endeavor Clinical Trials, San Antonio, Texas